CLINICAL TRIAL: NCT00924131
Title: Evaluation of Late Treatment Effects in Long-Term Survivors of Hodgkin's Disease Previously Treated at NIH: A Multi-Institutional Trial
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090127; 09-C-0127; NCT00909246 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-26

CONDITIONS: Hodgkin's Disease; Lymphoma
Keywords: Late Effects; Radiation; Chemotherapy; Hodgkin's Disease; Lymphoma; Hodgkin Disease
MeSH Terms: conditions — Hodgkin Disease; Lymphoma

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

* Researchers are greatly interested in knowing more about the long-term effects of various treatments for cancers such as Hodgkin's disease, particularly from those who have lived 20 to 30 years after treatment.
* Patients who were treated at the National Institutes of Health (NIH) may have undergone different treatments for which more long-term information is needed.

Objectives:

* To examine the body systems of long-term survivors of Hodgkin's disease to see if there are any long- term consequences of treatment for Hodgkin's disease.
* To learn more about the long-term effects of cancer treatments.

Eligibility:

* Survivors of Hodgkin's disease who were previously treated at the NIH.
* Participants must be at least 18 years of age.

Design:

* Participants will need to sign consent forms to allow researchers to obtain documentation of medical history, including prior treatment for Hodgkin's disease and prior NIH treatment, including protocol number, where applicable:
* Pertinent medical records, pathology reports, and radiographic imaging studies will be reviewed.
* Primary care physician's name, address, and other contact information are also required.
* Evaluations during the assessment period:
* Complete physical examination.
* Laboratory studies of blood, urine, and stool samples.
* Radiologic evaluations, including computerized tomography (CT) and magnetic resonance imaging (MRI) scans for all participants and mammograms for females.
* Cardiac evaluation, vascular studies, and pulmonary studies to measure heart and lung function, and digestive tests to measure stomach and intestinal function.
* Neurocognitive testing to measure brain function.
* Optional skin biopsy.
* Participants will be asked to complete questionnaires assessing current quality of life and daily living skills.

DETAILED DESCRIPTION:
BACKGROUND:

Nearly 75% of Hodgkin's Disease (HD) patients can be cured of their disease with chemotherapy and radiotherapy, resulting in a growing number of long-term survivors.

Adverse effects of HD treatments, including second malignancies and cardiovascular disease, affect survival and quality of life. Minimizing late toxicities has become a major emphasis of current and investigational regimens.

Better characterization of long-term toxicity and quality of life (QOL) after therapy for HD and the ability to determine which late toxicities arise from a given modality may allow an ability to shape future regimens such that late toxicity can be minimized.

OBJECTIVES:

Primary objectives:

To describe the cardiac, pulmonary, and vascular function in patients previously treated for HD at NIH and to correlate this information to the treatment received.

* To measure cardiac function and abnormalities and to correlate these findings with treatment received.
* To measure pulmonary function with pulmonary function testing in survivors of HD and to correlate these findings with treatment received.
* To measure vascular function in survivors of HD and to correlate these findings with treatment received.

Secondary Objectives:

To determine if elevated plasma TGF levels correlate with the presence of late radiation fibrosis in long-term survivors of HD.

To evaluate late quality of life (QOL) in long-term survivors of HD and to correlate QOL with treatment received.

To evaluate and describe additional exploratory measures of organ function in patients previously treated for HD at NIH and to correlate this information to the treatment received.

* Heart rate variability
* Pulmonary fibrosis.
* Intestinal function.
* Neurocognitive function.

To evaluate the correlation of exploratory functional assays, biomarkers, and single nucleotide polymorphisms with the presence of late chemotherapy or radiation toxicity in long-term HD survivors.

ELIGIBILITY:

Survivors of HD previously treated at the NIH.

DESIGN:

This is a single point in time follow-up evaluation of long-term HD survivors, previously treated at the NIH.

Patients will be evaluated for late toxicities in multiple organ systems using imaging modalities, laboratory tests, functional assays, and investigational studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for all Participants:

* Patients must be at least 18 years of age 15
* Patients must have been previously treated for Hodgkin's Disease at the NIH
* Patient must be willing to complete quality of life questionnaires and to answer questions regarding their medical history
* Patient must be willing to provide release of medical information forms for physicians and hospitals involved in their management

Inclusion Criteria for Evaluation at NIH/NIA:

In addition to those above,

* Patient is willing to return to NIH/NIA to participate in the protocol
* Patient must have a primary physician in the community who is willing to communicate with NIH regarding clinical findings and collaborate in the clinical management and follow-up of the patient. This will be substantiated by communicating directly with the patient's physician prior to evaluation.
* Pregnant patients are eligible for follow up evaluations and quality of life evaluations. They will be excluded for any radiological testing and invasive studies. Any blood draws will be approved by the patient's obstetrician and if any of the laboratory tests to be performed have been carried out within the last three months, those values will be used instead of repeating them. Alternatively, pregnant patients may choose to participate in the study after the birth of their child to be able to participate in the full evaluation.

EXCLUSION CRITERIA:

* Inability to give informed consent
* Patients, and/ or guardians who are in the estimation of the PI, deemed unable or unlikely to adhere to protocol evaluations and follow-up requirements.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2009-04-17; Study Completion 2010-05-26

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aisenberg AC. Problems in Hodgkin's disease management. Blood. 1999 Feb 1;93(3):761-79. No abstract available. PMID 9920825
- [Background] Fung HC, Nademanee AP. Approach to Hodgkin's lymphoma in the new millennium. Hematol Oncol. 2002 Mar;20(1):1-15. doi: 10.1002/hon.683. PMID 11921013
- [Background] AISENBERG AC. HODGKIN'S DISEASE--PROGNOSIS, TREATMENT AND ETIOLOGIC AND IMMUNOLOGIC CONSIDERATIONS. N Engl J Med. 1964 Mar 19;270:617-22 CONCL. doi: 10.1056/NEJM196403192701206. No abstract available. PMID 14096883